CLINICAL TRIAL: NCT00124020
Title: A Phase 3, Randomized, Double-Blind, Parallel-Group, Multinational Trial of Intravenous Telavancin Versus Vancomycin for Treatment of Hospital-Acquired Pneumonia With a Focus on Patients With Infections Due to Methicillin-Resistant Staphylococcus Aureus
Brief Title: Comparison of Telavancin and Vancomycin for Hospital-acquired Pneumonia Due to Methicillin-resistant Staphylococcus Aureus
Acronym: ATTAIN2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Steven L. Barriere, Pharm.D., Vice President, Clinical and Medical Affairs, Theravance, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0019
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Results first posted 2010-02-01 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2018-12

CONDITIONS: Bacterial Pneumonia
MeSH Terms: conditions — Pneumonia, Bacterial | interventions — telavancin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telavancin (Experimental)
  Interventions: Drug: Telavancin
- Vancomycin (Active Comparator)
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Telavancin — Telavancin 10 mg/kg/day IV for up to 21 days
  Other Names: TD6424; VIBATIV
  Arms: Telavancin
Drug: Vancomycin — Vancomycin 1 Gm administered every 12 hrs IV for up to 21 days
  Arms: Vancomycin

SUMMARY:
Study 0019 (NCT00124020) compares the safety and effectiveness of an investigational drug, telavancin, with vancomycin for the treatment of hospital-acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs and symptoms consistent with pneumonia acquired after at least 48 hours of continuous stay in an inpatient acute or chronic care facility or acquired within 7 days after being discharged from a hospitalization of greater than or equal to 3 days duration.

Exclusion Criteria:

* Received more than 24 hours of potentially effective systemic (IV, IM or PO) antibiotic therapy for Gram-positive pneumonia immediately prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 771 (Actual)
Dates: Start 2005-01; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G. Ralph Corey, MD, Principal Investigator — Duke University
Locations (1):
- Sheba Medical Center, Infectious Disease Unit, Tel Litwinsky, Israel

REFERENCES:
- [Derived] McKinnell JA, Corman S, Patel D, Leung GH, Gordon LM, Lodise TP. Effective Antimicrobial Stewardship Strategies for Cost-effective Utilization of Telavancin for the Treatment of Patients With Hospital-acquired Bacterial Pneumonia Caused by Staphylococcus aureus. Clin Ther. 2018 Mar;40(3):406-414.e2. doi: 10.1016/j.clinthera.2018.01.010. Epub 2018 Feb 15. PMID 29454592
- [Derived] Smart JI, Corey GR, Stryjewski ME, Wang W, Barriere SL. Assessment of Minimum Inhibitory Concentrations of Telavancin by Revised Broth Microdilution Method in Phase 3 Hospital-Acquired Pneumonia/Ventilator-Associated Pneumonia Clinical Isolates. Infect Dis Ther. 2016 Dec;5(4):535-544. doi: 10.1007/s40121-016-0133-y. Epub 2016 Oct 7. PMID 27718118
- [Derived] Barriere SL, Stryjewski ME, Corey GR, Genter FC, Rubinstein E. Effect of vancomycin serum trough levels on outcomes in patients with nosocomial pneumonia due to Staphylococcus aureus: a retrospective, post hoc, subgroup analysis of the Phase 3 ATTAIN studies. BMC Infect Dis. 2014 Apr 4;14:183. doi: 10.1186/1471-2334-14-183. PMID 24708675

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Period: 23 January 2005 to 02 May 2007
Pre-assignment Details: 14 patients (9 telavancin and 5 vancomycin) enrolled in the study but never started study treatment
Groups:
- Telavancin: Patients with Gram-positive hospital acquired pneumonia (HAP) (primarily due to MRSA) were randomized to receive telavancin 10 mg/kg IV every 24 hrs
- Vancomycin: Patients with Gram-positive hospital acquired pneumonia (HAP)(primarily due to MRSA) were randomized to receive vancomycin 1 Gm IV every 12 hrs.
Period: Overall Study
Arm/Group | Telavancin | Vancomycin
Started | 377 | 380
Completed | 289 | 289
Not Completed | 88 | 91
Not completed — Death | 67 | 71
Not completed — Withdrawal by Subject | 13 | 11
Not completed — Lost to Follow-up | 5 | 8
Not completed — Other | 1 | 1
Not completed — Transfer to another hospital | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telavancin | Vancomycin | Total
Number analyzed (Participants) | 377 | 380 | 757
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 182 | 184 | 366
  >=65 years | 195 | 196 | 391
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (17.8) | 62 (18.0) | 62 (17.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 124 | 249
  Male | 252 | 256 | 508
Region of Enrollment [Number; unit: participants]
  Argentina | 20 | 19 | 39
  Australia | 9 | 14 | 23
  Brazil | 17 | 16 | 33
  Bulgaria | 20 | 20 | 40
  Canada | 3 | 10 | 13
  Chile | 0 | 5 | 5
  China | 27 | 37 | 64
  Croatia | 2 | 2 | 4
  Czech Republic | 3 | 1 | 4
  Estonia | 0 | 1 | 1
  France | 1 | 1 | 2
  Georgia | 17 | 13 | 30
  Greece | 1 | 1 | 2
  Israel | 38 | 38 | 76
  Korea, Republic of | 23 | 30 | 53
  Lebanon | 5 | 4 | 9
  Lithuania | 7 | 10 | 17
  Mexico | 31 | 29 | 60
  Philippines | 8 | 9 | 17
  Poland | 6 | 4 | 10
  Romania | 4 | 3 | 7
  Russian Federation | 21 | 29 | 50
  Serbia | 7 | 10 | 17
  Slovakia | 6 | 6 | 12
  South Africa | 7 | 3 | 10
  Spain | 0 | 2 | 2
  Thailand | 22 | 11 | 33
  Ukraine | 12 | 6 | 18
  United States | 60 | 46 | 106
Diabetes Status [Number; unit: participants]
  Diabetic | 69 | 65 | 134
  Non-Diabetic | 308 | 315 | 623
History of Pneumonia [Number; unit: participants]
  Prior history of pneumonia | 37 | 45 | 82
  No prior history of pneumonia | 340 | 335 | 675
Ventilator Status [Number; unit: participants]
  Ventilated | 175 | 175 | 350
  Non-ventilated | 202 | 205 | 407

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: Clinical Response: Categorical (Cured, Failed or Indeterminate)
  * Failure - at least one of the following:
  * Persistence or progression of signs and symptoms of pneumonia that still require antibiotic therapy
  * Termination of study med due to "lack of efficacy"
  * Death on or after Day 3 attributable to primary infection
  * Cure: Signs and symptoms of pneumonia improved to the point that no further antibiotics for pneumonia were required, and baseline radiographic findings improved or did not progress.
  * Indeterminate: Inability to determine outcome
Time Frame: 7-14 days following end of antibiotic treatment
Measure: Number; unit: participants
Arm/Group | Telavancin | Vancomycin
Number analyzed (Participants) | 377 | 380
participants
  Cured | 227 | 228
  Failure | 53 | 52
  Indeterminate | 39 | 38
  Missing | 58 | 62
Statistical Analysis 1: Comparison: Telavancin vs Vancomycin; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 20% was specified based on historical regulatory precedent; p-values were not calculated in deference to confidence intervals; Risk Difference (RD) = 0.2, 95% CI [-6.8 to 7.2]

ADVERSE EVENTS:
Description: Two patients were randomized to vancomycin, yet were treated with telavancin. For analyses of efficacy, results were analyzed according to the treatment group assigned by randomization. For safety analyses, results were analyzed according to treatment received; 379 patients received telavancin and 378 patients received vancomycin.
Arm/Group | Telavancin | Vancomycin
Serious Adverse Events (participants affected / at risk) | 107/379 | 109/378
Other Adverse Events (participants affected / at risk) | 295/379 | 296/378
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telavancin (N=379) | Vancomycin (N=378)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 2
Bradycardia (Cardiac disorders) | 0 | 2
Cardiac Arrest (Cardiac disorders) | 5 | 0
Cardiac failure (Cardiac disorders) | 1 | 3
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 7
Cardiogenic Shock (Cardiac disorders) | 1 | 2
Cardiopulmonary Failure (Cardiac disorders) | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Wandering pacemaker (Cardiac disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 | 0
Gastrointestinal Necrosis (Gastrointestinal disorders) | 0 | 1
Mesenteric Occlusion (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 2
Multi-organ Failure (General disorders) | 13 | 6
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Hepatocellular damage (Hepatobiliary disorders) | 0 | 1
Abdominal Abscess (Infections and infestations) | 1 | 0
Abdominal Sepsis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial Sepsis (Infections and infestations) | 1 | 0
Candida Sepsis (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Lung Infection pseudomonal (Infections and infestations) | 2 | 0
Meningitis (Infections and infestations) | 3 | 2
Meningitis Candida (Infections and infestations) | 0 | 1
Peritonitis Bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 6
Pneumonia Staphylococcal (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 6 | 5
Septic Shock (Infections and infestations) | 17 | 15
Sinusitis fungal (Infections and infestations) | 1 | 0
Superinfection Lung (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 0 | 2
Urosepsis (Infections and infestations) | 0 | 1
Anastomotic Stenosis (Injury, poisoning and procedural complications) | 0 | 1
Brain herniation (Injury, poisoning and procedural complications) | 1 | 0
Post-operative ileus (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1
Wound Evisceration (Injury, poisoning and procedural complications) | 1 | 0
Blood Potassium increased (Investigations) | 0 | 1
Blood sodium increased (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Bile Duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small Cell Lung Cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 1
Cerebellar Haemorrhage (Nervous system disorders) | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1
Cerebral ischemia (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 4 | 3
Convulsion (Nervous system disorders) | 0 | 2
Dementia (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Intracranial Pressure increased (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 0
Neurological Symptom (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 7 | 8
Renal Failure Chronic (Renal and urinary disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 1
Renal Insufficiency (Renal and urinary disorders) | 1 | 0
Urine flow decreased (Renal and urinary disorders) | 1 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Airways Disease Exacerbated (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax Spontaneous Tension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pulmonary Necrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Throat secretion increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arterial Rupture (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 0 | 3
Shock (Vascular disorders) | 3 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telavancin (N=379) | Vancomycin (N=378)
Anemia (Blood and lymphatic system disorders) | 34 | 36
Leukocytosis (Blood and lymphatic system disorders) | 11 | 9
Thrombocythaemia (Blood and lymphatic system disorders) | 4 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 7
Atrial fibrillation (Cardiac disorders) | 15 | 18
Bradycardia (Cardiac disorders) | 5 | 6
Cardiac failure (Cardiac disorders) | 3 | 7
Cardiac failure congestive (Cardiac disorders) | 9 | 12
Tachycardia (Cardiac disorders) | 12 | 7
Ventricular Extrasystoles (Cardiac disorders) | 5 | 7
Ventricular tachycardia (Cardiac disorders) | 0 | 7
Abdominal distension (Gastrointestinal disorders) | 7 | 5
Abdominal Pain (Gastrointestinal disorders) | 4 | 11
Constipation (Gastrointestinal disorders) | 38 | 35
Diarrhoea (Gastrointestinal disorders) | 38 | 38
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 8 | 12
Nausea (Gastrointestinal disorders) | 13 | 12
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 | 7
Vomiting (Gastrointestinal disorders) | 15 | 12
Anasarca (General disorders) | 7 | 8
Multi-organ Failure (General disorders) | 13 | 6
Oedema Peripheral (General disorders) | 14 | 12
Pain (General disorders) | 3 | 6
Bacteraemia (Infections and infestations) | 6 | 2
Oral Candidiasis (Infections and infestations) | 5 | 6
Pneumonia (Infections and infestations) | 8 | 7
Sepsis (Infections and infestations) | 17 | 7
Septic Shock (Infections and infestations) | 17 | 16
Urinary Tract Infection (Infections and infestations) | 14 | 9
Post-Procedural Haemorrhage (Injury, poisoning and procedural complications) | 4 | 6
Post-Procedural Pain (Injury, poisoning and procedural complications) | 4 | 6
Alanine Aminotransferase increased (Investigations) | 10 | 17
Aspartate Aminotransferase increased (Investigations) | 10 | 13
Blood Creatinine Increased (Investigations) | 7 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 16 | 17
Hyperkalaemia (Metabolism and nutrition disorders) | 13 | 10
Hypernatremia (Metabolism and nutrition disorders) | 6 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 14 | 9
Hypokalemia (Metabolism and nutrition disorders) | 31 | 39
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 7
Hyponatremia (Metabolism and nutrition disorders) | 8 | 11
Malnutrition (Metabolism and nutrition disorders) | 6 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 7 | 4
Convulsion (Nervous system disorders) | 5 | 9
Headache (Nervous system disorders) | 13 | 10
Agitation (Psychiatric disorders) | 8 | 11
Anxiety (Psychiatric disorders) | 12 | 12
Confusional State (Psychiatric disorders) | 3 | 7
Depression (Psychiatric disorders) | 9 | 3
Insomnia (Psychiatric disorders) | 18 | 15
Renal Failure Acute (Renal and urinary disorders) | 16 | 18
Renal Impairment (Renal and urinary disorders) | 6 | 4
Renal Insufficiency (Renal and urinary disorders) | 7 | 3
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Dependence on Respirator (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Decubitis Ulcer (Skin and subcutaneous tissue disorders) | 17 | 18
Erythema (Skin and subcutaneous tissue disorders) | 7 | 7
Rash (Skin and subcutaneous tissue disorders) | 12 | 16
Hypertension (Vascular disorders) | 21 | 12
Hypotension (Vascular disorders) | 25 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less